CLINICAL TRIAL: NCT04718935
Title: Nutritional and Metabolic Biomarkers in Prediction of Outcomes After Traumatic Brain Injury: a Patient Cohort Study
Acronym: PATOSTBI
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other); SMG-SNU Boramae Medical Center (Other); Kyungpook National University Hospital (Other); Chonnam National University Hospital (Other); Chungbuk National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SNUEMSTBI21
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-04

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — To investigate biomarkers, 20ml of blood is collected from study subjects. Blood is collected first in 2 SST tubes that do not contain anticoagulant, and then blood is collected in 1 EDTA tube containing anticoagulant. Leave blood sample at room temperature for 1 hour and then centrifuge for 10 minutes. Finally, the sample separated by serum, plasma, and buffy coat is stored frozen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To identify nutritional and metabolic biomarkers that are related to the prognosis of traumatic brain injury patients, and to develop a prognosis prediction model using biomarkers

Study Objectives:

1. Establishment of a prospective registry for traumatic brain injury patients
2. Identification of nutritional and metabolic biomarkers related to prognosis of traumatic brain injury patients
3. Development of a prognosis prediction model using nutritional and metabolic biomarkers
4. Development of identification model for high-risk population of disabilities after traumatic brain injury

DETAILED DESCRIPTION:
Study design: Multicenter observational cohort study, 5 tertiary teaching hospital emergency departments in Korea

Study period: July 2018 to December 2023 (66 months)

Study population: Traumatic brain injury patients aged over 18.

Cases will be consecutive adult patients with EMS-treated traumatic brain injury and transport to the 5 emergency departments of participating hospitals within 72 hours after the trauma and confirmed cerebral hemorrhage or diffuse axial injury by radiological examination. A prospective traumatic brain injury patient cohort will be developed and all survived traumatic brain injury cases will be followed at 1-month and 6-month after ED discharge by telephone.

During the study period, the investigators aim to recruit a total 1,200 cases (600 cases between July 2018 and June 2020, 600 cases between March 2021 and June 2023).

Data collection: Following data will be collected

Clinical data: Basic demographic and clinical outcomes will be retrieved from medical records.

Survey data: Comorbidity, symptom, result of neurologic examination, socioeconomic status (occupation, income etc) data will be collected.

Blood samples: The investigators aim to develop nutritional and metabolic biomarkers of traumatic brain injury. The investigators also plan to further develop traumatic brain injury biomarkers using proteomics.

Follow-ups: All survived traumatic brain injury cases will be followed-up at 1-month and 6-month after ED discharge and their survival, disability, and quality of life outcomes will be collected by telephone.

Ethics Statements: All 5 hospitals participating in the study were IRB approved(Seoul National University Hospital(IRB No: 1806-078-951), SMG-SNU Boramae Medical Center(IRB No: 30-2018-85), Kyungpook National University Hospital(IRB No: 2018-10-014-007), Chonnam National University Hospital(IRB No: CNUH-2018-297), Chungbuk National University Hospital(IRB No: 2018-09-018)). All study patients was registered in cohort after acquisition of consent.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years old
* Traumatic brain injury patient transported by EMS ambulance to the emergency department of the participating hospital or transporting from another hospital emergency room (EMS treated traumatic brain injury)
* Visiting emergency department of the participating hospital within 72 hours after trauma
* With confirmed intracranial damage such as cerebral hemorrhage or diffuse axial injury by imaging

Exclusion Criteria:

* People who do not consent to personal information and blood supply for research.
* With penetrating brain injury
* Patients with known neurological disease, psychiatric disorder.
* Pregnant patient
* Patients with a terminal condition known to have no further treatment plans due to malignancy. The terminal condition had to be checked by a doctor or recorded in medical records.
* Patients who were transported after surgery at the other hospital.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases will be consecutive adult patients with EMS-treated traumatic brain injury and transport to the 5 emergency departments of participating hospitals.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Survival of traumatic brain injury patient | 6 months after traumatic brain injury
  survival, cause of death
Functional outcome of traumatic brain injury patient | 6 months after traumatic brain injury
  Glasgow Outcome Scale
Quality of life of traumatic brain injury patient | 6 months after traumatic brain injury
  EQ-5D

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No